CLINICAL TRIAL: NCT07172412
Title: An Umbrella Ib/II Phase Study Evaluating the Efficacy and Safety of First-Line Combination Therapy in the Treatment of Extensive-Stage Small Cell Lung Cancer
Brief Title: Open-Label, Biomarker-Integrated Umbrella Trial for First-Line Treatment of Extensive-stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BUTTONS-001
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Extensive Stage Lung Small Cell Cancer
MeSH Terms: interventions — selinexor; anlotinib; Etoposide; Cisplatin; Carboplatin; tislelizumab; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anlotinib TEAM (Experimental): Anlotinib+SOC therapy
  Interventions: Drug: Anlotinib; Drug: Etoposide + Cisplatin/Carboplatin; Drug: Tislelizumab/Atezolizumab/ Durvalumab/Benmelstobart/Toripalimab/Serplulimab
- DLL3 TEAM (Experimental): DLL3 CAR-NK cell+SOC therapy
  Interventions: Biological: DLL3 CAR-NK cells; Drug: Etoposide + Cisplatin/Carboplatin; Drug: Tislelizumab/Atezolizumab/ Durvalumab/Benmelstobart/Toripalimab/Serplulimab
- XPO1 TEAM (Experimental): Selinexor+SOC therapy
  Interventions: Drug: Selinexor; Drug: Etoposide + Cisplatin/Carboplatin; Drug: Tislelizumab/Atezolizumab/ Durvalumab/Benmelstobart/Toripalimab/Serplulimab

INTERVENTIONS:
Drug: Selinexor — Selinexor 60 mg biw q21d
  Arms: XPO1 TEAM
Drug: Anlotinib — Anlotinib 12mg d1-14 qd PO
  Arms: Anlotinib TEAM
Biological: DLL3 CAR-NK cells — 1.0×10^9 DLL3-CAR-NK+ cells d5 q6w
  Arms: DLL3 TEAM
Drug: Etoposide + Cisplatin/Carboplatin — Etoposide 100mg/m^2 d1-3+ cisplatin 75mg/m^2 d1-3 or Carboplatin AUC5
Drug: Tislelizumab/Atezolizumab/ Durvalumab/Benmelstobart/Toripalimab/Serplulimab — Use immunotherapy according to the standard immunotherapy-combined-chemotherapy protocol.

SUMMARY:
This is an open-label umbrella study conducted in first treatment ES-SCLC patients, employing a novel umbrella trial design (biomarker-integrated multi-arm trial with a shared ICI+chemotherapy control arm). Eligible patients were assigned to trial arms based on biomarker expression levels. Biomarker subgroups were defined as: (1) High ASCL1/NEUROD1/DLL3 expression: DLL3-CAR-NK cells combined with ICI + etoposide + carboplatin (DLL3 group); (2) Myc overexpression: XPO1 inhibitor selinexor combined with ICI + etoposide + carboplatin (XPO1 group); (3) VIM/AXL high expression group treated with anlotinib combined with ICI + etoposide + carboplatin (anlotinib group).

DETAILED DESCRIPTION:
Patients received specific targeted therapy combined with SOC treatment (etoposide 100 mg/m² on days 1-3 + carboplatin AUC5 on day 1 + immunotherapy on day 1): (1) DLL3 cohort: 1.0 × 10^9 DLL3-CAR-positive NK cells d5 q6w; (2) XPO1 cohort: Oral selinexor 60 mg biweekly q21d; (3) Anlotinib cohort: Oral anlotinib 12 mg on days 1-14, q21d.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of SCLC is confirmed by histology or cytology, and according to VALSG and AJCC9, the imaging diagnosis is extensive stage.
* Patients who have not previously received systemic therapy for advanced or metastatic disease, or patients who have relapsed after concurrent chemo-radiotherapy during the localized stage.
* The expected survival time is not less than 12 weeks.
* According to RECIST V1.1, there is at least one measurable lesion that has not undergone radiation therapy.
* The Eastern Cooperative Oncology Group (ECOG) physical condition score is evaluated as 0 or 1.
* When screening, there is sufficient bone marrow reserve, and no blood transfusion or hematopoietic stimulating factor treatment has been received 10 days before the test. The definition is as follows: absolute neutrophil counts (ANC) ≥ 1.5×109/L, platelet (PLT) ≥ 100×109/L and hemoglobin (HGB) ≥ 90g/L.
* Appropriate organ function during screening, meeting the following criteria: aspartate aminotransferase (AST) ≤ 2.5×ULN (with liver metastasis ≤ 5×ULN); alanine aminotransferase (ALT) ≤ 2.5ULN (with liver metastasis ≤ 5ULN); total serum bilirubin ≤ 1.5×ULN (with tumor infiltration ≤ 3×ULN); serum creatinine (Scr) ≤ 1.5×ULN, or creatinine clearance rate ≥ 60mL/min; international normalized ratio (INR) ≤ 1.5×ULN, and activated partial thromboplastin time (APTT) ≤ 1.5×ULN; the urine pregnancy test for women of childbearing age needs to be negative, and any male and female patients with fertility must agree to use effective contraceptive methods throughout the entire study process and for at least 1 year after treatment.

Exclusion Criteria:

* During screening, patients with symptomatic central nervous system (CNS) metastasis (asymptomatic CNS metastasis, or asymptomatic and stable condition after local treatment for 4 weeks can be enrolled).
* Individuals with a history of central nervous system diseases before screening, such as epilepsy, cerebral ischemia/bleeding, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, mental illness, or any autoimmune disease associated with central nervous system involvement.
* Received chemotherapy, radiation therapy, immunotherapy, targeted therapy, biological therapy, endocrine therapy within 4 weeks of screening, and was evaluated by the researcher as not suitable for enrollment.
* The adverse reactions of previous anti-tumor treatments have not yet recovered to level 1 (CTCAE5.0), except for toxicity that the researchers have determined to have no safety risk, such as hair loss and level 2 peripheral neurotoxicity.
* Those who discontinue systemic hormone therapy for less than 72 hours before the first administration, but are allowed to use physiological replacement doses of hormones (such as prednisone < 10mg/d or equivalent).
* Received organ/tissue transplantation before screening.
* Prior to screening, it was known that the patient had active systemic autoimmune diseases and was currently undergoing treatment.
* Those who meet any of the following conditions during screening: hepatitis B surface antigen (HBsAg) is positive, and the copy number of HBV DNA is greater than the measurable lower limit; hepatitis C antibody (HCV Ab) is positive; treponema pallidum antibody (TP-Ab) is positive; HIV antibody is positive; The copy numbers of EBV-DNA and CMV-DNA are higher than the measurable lower limit.
* Individuals who have undergone major surgery or experienced significant trauma within 4 weeks prior to screening, or who require elective surgery during the trial period, have been evaluated by the researchers as unsuitable for inclusion.
* Within 2 years prior to screening or currently suffering from other malignant tumors.
* When screening, the heart meets any of the following conditions: New York Heart Association (NYHA) ≥ Level II, Left Ventricular Ejection Fraction (LVEF) ≤ 50% (ECHO); Hypertension (systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg) or pulmonary hypertension that has not been controlled after standardized treatment; Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other Grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before the first administration; valvular disease with clinical significance; There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias that require clinical intervention, II-III degree atrioventricular block, etc.
* Patients with tumor involving the atrium or ventricle during screening.
* When screening, there are clinical emergencies that require urgent treatment due to tumor obstruction or compression (such as intestinal obstruction or vascular compression).
* Individuals with active bleeding during screening.
* Those with a history of deep vein thrombosis or pulmonary embolism within 6 months before screening.
* Individuals who have received live vaccines within 6 weeks before screening.
* Subjects with uncontrolled systemic bacterial, viral, or fungal infections after optimal treatment.
* Participated in other interventional clinical studies within 4 weeks before the first administration.
* Individuals with poor adherence or those who are deemed unsuitable for clinical trials by researchers due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 1 year
ORR | through study completion, an average of 1 year
OS | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China 300060, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion

REFERENCES:
- [Background] Liu Q, Zhang J, Guo C, Wang M, Wang C, Yan Y, Sun L, Wang D, Zhang L, Yu H, Hou L, Wu C, Zhu Y, Jiang G, Zhu H, Zhou Y, Fang S, Zhang T, Hu L, Li J, Liu Y, Zhang H, Zhang B, Ding L, Robles AI, Rodriguez H, Gao D, Ji H, Zhou H, Zhang P. Proteogenomic characterization of small cell lung cancer identifies biological insights and subtype-specific therapeutic strategies. Cell. 2024 Jan 4;187(1):184-203.e28. doi: 10.1016/j.cell.2023.12.004. PMID 38181741
- [Background] Wang J, Sun T, Meng Z, Wang L, Li M, Chen J, Qin T, Yu J, Zhang M, Bie Z, Dong Z, Jiang X, Lin L, Zhang C, Liu Z, Jiang R, Yang G, Li L, Zhang Y, Huang D. XPO1 inhibition synergizes with PARP1 inhibition in small cell lung cancer by targeting nuclear transport of FOXO3a. Cancer Lett. 2021 Apr 10;503:197-212. doi: 10.1016/j.canlet.2021.01.008. Epub 2021 Jan 23. PMID 33493586
- [Background] Qin T, Wang J, Wang J, Du Q, Wang L, Liu H, Liu W, Li X, Jiang Y, Xu Q, Yu J, Liu H, Wang T, Li M, Huang D. Nuclear to Cytoplasmic Transport Is a Druggable Dependency in HDAC7-driven Small Cell Lung Cancer. Adv Sci (Weinh). 2025 Apr;12(14):e2413445. doi: 10.1002/advs.202413445. Epub 2025 Jan 30. PMID 39887933